CLINICAL TRIAL: NCT03018808
Title: A Cross-sectional Study to Characterize the Prevalence of COPD and Eosinophilia Among Primary Care Patients in Brazil
Brief Title: Prevalence of Chronic Obstructive Pulmonary Disease (COPD) and Eosinophilia Among Primary Care Patients
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 207620
Record Dates: First submitted 2017-01-10; First posted 2017-01-12 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Eosinophilia; COPD prevalence; Primary care subjects
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Eosinophilia | interventions — Hematologic Tests; Oximetry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Subjects met inclusion with at least one exclusion criteria: Subjects who meet all the inclusion criteria, but have at least one exclusion criteria or not agree to participate in the whole study will be invited to sign a special ICF in order to complete a minimal questionnaire.
  Interventions: Other: Minimal questionnaire; Other: CAT; Procedure: Blood test; Other: anthropometric measures; Other: Oximetry
- Subjects who satisfy all inclusion/exclusion criteria: Subjects who satisfy all inclusion/exclusion criteria and agree to sign the ICF, an interview will be conducted for information regarding medical history, sociodemographic and clinical information, including disease history, treatment history, smoking habits and use of biomass.
  Interventions: Other: Medical interview; Other: CAT; Procedure: Blood test; Other: anthropometric measures; Other: Oximetry
- Spirometry confirmed COPD Subjects: The spirometry confirmed COPD patients will be requested to complete the COPD Assessment Test (CAT), self-administered questionnaire related to quality of life on COPD patients.
  Interventions: Other: Medical interview; Other: CAT

INTERVENTIONS:
Other: Minimal questionnaire — The minimal questionnaire is a reduced version of the medical interview and it will include questions about sociodemographic information, previous diagnosis of COPD, co-morbidities and smoking habits.
  Groups: Subjects met inclusion with at least one exclusion criteria
Other: Medical interview — Medical interview includes medical history, sociodemographic and clinical information, including disease history, treatment history, smoking habits and use of biomass.
  Groups: Spirometry confirmed COPD Subjects; Subjects who satisfy all inclusion/exclusion criteria
Other: CAT — The CAT is a questionnaire for COPD patients and is designed to measure the impact of COPD on a person's life over time.
Procedure: Blood test — Blood samples will be collected at indicated time points
  Groups: Subjects met inclusion with at least one exclusion criteria; Subjects who satisfy all inclusion/exclusion criteria
Other: anthropometric measures — Anthropologic measures will be performed.
  Groups: Subjects met inclusion with at least one exclusion criteria; Subjects who satisfy all inclusion/exclusion criteria
Other: Oximetry — Digital pulse oximeter on the index finger after five minutes rest and before receiving bronchodilator for spirometry will be used to measure the pulse arterial oximetry. The average of three measurements at 10 second intervals will be recorded. The heart rate will be provided by the pulse oximeter.
  Groups: Subjects met inclusion with at least one exclusion criteria; Subjects who satisfy all inclusion/exclusion criteria

SUMMARY:
Early diagnosis and appropriate treatment for COPD subjects are both critical to minimize the progression of COPD and improve outcomes. Also, evidence suggests that high eosinophil (specific type of white blood cell that protects body against certain kinds of germs) level is associated with increased risk of both moderate and severe exacerbations in COPD subjects. To date, there is insufficient amount of data that describes the prevalence of COPD in Brazilian primary care units. Thus, this multicenter, cross-sectional study conducted in five centers located in five different Brazilian cities will provide estimation about the prevalence of COPD in primary care and will also determine the levels of eosinophils in subjects with confirmed COPD diagnosis. Approximately 2,500 eligible subjects are expected to be enrolled in the study.

DETAILED DESCRIPTION:
The study is a cross sectional (prevalence study).

ELIGIBILITY:
Inclusion Criteria:

* Adult >= 35 years old
* At least one of the following risk factors for COPD:

  • being a current smoker (who has smoked 100 cigarettes in his or her lifetime and who currently smokes cigarettes) or past smoker (who has smoked at least 100 cigarettes in his or her lifetime but who had quit smoking at the time of interview); Current or past exposure to biomass smoke, such as wood or coal, for cooking or heating (exposure >=100 hours/year
* Capable of giving signed informed consent

Exclusion Criteria:

* Physical or mental disability to complete the study procedures
* Heart above 120 beats per minute
* Participants under treatment for tuberculosis
* Participant in current clinical trial
* Pregnancy
* Patients with one of the following contraindications to spirometry: chest surgery in the last month; abdominal surgery within the past three months; neuromuscular disease, acute coronary syndrome; retinal detachment; hospitalization for any cardiac problem in the prior 3 months.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects over 35 years, with at least one COPD risk factor, who visit the Basic Health Unit (BHU) for a routine, spontaneous or scheduled medical visit for any cause
Sampling Method: Probability Sample
Enrollment: 800 (Actual)
Dates: Start 2019-06-03 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
Number of subjects with spirometry confirmed COPD diagnosis according to Fixed Ratio Criteria | Day 1
  Spirometry confirmed COPD diagnosis according to fixed ratio criteria will be defined as those with post-Bronchodilatador (BD) Forced Expiratory Volume in 1 second (FEV1)/ Forced Vital Capacity (FVC) < 0.7 among the total of patients with valid spirometry. Spirometry tests will be performed at Baseline and 15 minutes after the administration of 400 microgram (mcg) Salbutamol.
Number of subjects with spirometry confirmed COPD diagnosis according to Lower Limit of Normal (LLN) Criteria | Day 1
  Spirometry confirmed COPD diagnosis according to Lower limit of normal (LNN) criteria will be defined as those with lower 5th percentile for predicted post-BD FEV1/FVC Spirometry tests will be performed at Baseline and 15 minutes after the administration of 400 mcg Salbutamol.
Number of subjects who self-reported physician diagnosis of COPD | Day 1
  Number of subjects that self-report physician diagnosis of emphysema, chronic bronchitis, or COPD.
Number of subjects with under diagnosed COPD | Day 1
  Number of subjects who meet the spirometry confirmed criteria of COPD (post-BD FEV1/FVC<0.7) but do not self-report medical diagnosis of emphysema, chronic bronchitis, or COPD.
Number of subjects with physician COPD diagnosis | Day 1
  Number of subjects who meet the spirometry confirmed criteria of COPD(post-BD FEV1/FVC<0.7) and self-report medical diagnosis of emphysema, chronic bronchitis, or COPD.
Number of subjects with misdiagnosed COPD | Day 1
  Number of subjects who do not meet the spirometry confirmed criteria of COPD but self-report diagnosis of emphysema, chronic bronchitis, or COPD.

SECONDARY OUTCOMES:
Number OF COPD subjects classified by Global Initiative for Chronic Obstructive Lung Disease (GOLD) Severity Groups | Day 1
  COPD subjects will be classified using the following severity classification: GOLD 2007 (GOLD, 2007); GOLD 2013 (GOLD, 2013); GOLD 2017 (GOLD, 2017).
Mean Charlson Comorbidity Index (CCI) score | Day 1
  All comorbidities included in the CCI will be investigated. The CCI contains 19 categories of comorbidity and predicts the ten-year mortality for a subject who may have a range of co-morbid conditions.
Descriptive statistics for COPD Assessment Test (CAT) score | Day 1
  Mean, Median, Max-Min, Q1-Q3 for CAT score will be described.
Number of subjects with mild exacerbation | Day 1
  Mild exacerbation will be defined as the deterioration of breathing symptoms that affected usual daily activities self-reported by the subject.
Number of subjects moderate exacerbation | Day 1
  Moderate exacerbation will be defined as the one for which subjects need to take antibiotic and/or systemic corticosteroid due to increase of cough, phlegm or breathlessness.
Number of subjects with severe exacerbation | Day 1
  Proportion of patients that needed to be hospitalized due to increase of cough, phlegm or breathlessness
Assessment of treatment used in the last 14 days and an last year | Day 1
  Subjects will report the COPD medication used in the last 14 days and in the last year.
Type of access to treatment | Day 1
  Subject will report where the medication (s) were obtained from (Public Health System, commercial pharmacy, charity institution/church, Brazilian Popular Pharmacy Program, free sample, friends/family/neighbor or other) at the last time they need such medication.
Number of subjects with Asthma-COPD Overlap (ACO) | Day 1
  It will be considered two definitions for considering a patient with ACO: 1) Subjects with Spirometry confirmed COPD post- BD increase in FEV1 or FVC of 200 milliliter (mL) and 12 percent plus self-reported wheezing in the last 12 months reported on the medical interview among all subjects with spirometry confirmed COPD. 2) subjects having a spirometry confirmed COPD and self-reported asthma physician diagnosis among all subjects with spirometry confirmed COPD.
Descriptive statistics for blood eosinophil's concentration | Day 1
  Geometric mean accompanied with 95% confidence intervals
Number of subjects with blood eosinophil's < 150, >= 150; <300 and >= 300 Cells/Microliter | Day 1
  A 5 mL sample of venous blood will be collected from each subject in order to have the complete blood count with differential count.
Number of subjects classified by Brazilian Society of Pulmonology and Physiology (SBPT) severity groups | Day 1
  COPD subjects will be classified using the SBPT 2017 classification system.
Descriptive statistics for FEV1 | Day 1
  Descriptive statistics for FEV1 will be summarized.
Mean CCI score as a measure of clinical characteristics by ACO definitions | Day 1
  All comorbidities included in the CCI will be investigated. The CCI contains 19 categories of comorbidity and predicts the ten-year mortality for a subject who may have a range of co-morbid conditions. Each condition is assigned a score of 1, 2, 3, or 6, depending on the risk of dying associated with each one.
Descriptive statistics for CAT score as a measure of clinical characteristics by ACO definitions | Day 1
  Mean, Median, Max-Min, Q1-Q3 for CAT score will be described.
Descriptive statistics for FEV1 as a measure of clinical characteristics by ACO definitions | Day 1
  Descriptive statistics for FEV1 will be summarized.
Number of subjects with mild exacerbation by ACO definition | Day 1
  Mild Exacerbation will be defined as the deterioration of breathing symptoms that affected usual daily activities self-reported by the subject.
Number of subjects with moderate exacerbation by ACO definition | Day 1
  Moderate exacerbation will be defined as the one for which subjects need to take antibiotic and/or systemic corticosteroid due to increase of cough, phlegm or breathlessness.
Number of subjects with severe exacerbation by ACO definition | Day 1
  Proportion of patients that needed to be hospitalized due to increase of cough, phlegm or breathlessness.
Mean CCI score as a measure of clinical characteristics of eosinophil groups | Day 1
  All comorbidities included in the CCI will be investigated. The CCI contains 19 categories of comorbidity and predicts the ten-year mortality for a subject who may have a range of co-morbid conditions.
Descriptive statistics for CAT score as a measure of clinical characteristics of eosinophil groups | Day 1
  Mean, Median, Max-Min, Q1-Q3 for CAT score will be described. Subjects identified with COPD will complete the CAT to measure the impact of COPD on a person's life.
Descriptive statistics for FEV1 as a measure of clinical characteristics of eosinophil groups | Day 1
  Descriptive statistics for FEV1 will be summarized.
Number of subjects with mild exacerbation of eosinophil groups | Day 1
  Mild Exacerbation will be defined as the deterioration of breathing symptoms that affected usual daily activities self-reported by the subject.
Number of subjects with moderate exacerbation of eosinophil groups | Day 1
  Moderate exacerbation will be defined as the one for which subjects need to take antibiotic and/or systemic corticosteroid due to increase of cough, phlegm or breathlessness.
Number of subjects with severe exacerbation of eosinophil groups | Day 1
  Proportion of patients that needed to be hospitalized due to increase of cough, phlegm or breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Brazil (4):
  - GSK Investigational Site, Londrina, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Araraquara, São Paulo
  - GSK Investigational Site, Botucatu, São Paulo